CLINICAL TRIAL: NCT01400061
Title: Phase 1 Study of Blood Boron Levels According to Body Mas Index
Brief Title: Relation of Blood-boron Levels With Body Mass Index
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Bezmialem Vakif University, bezmialem vakif university
Other Study IDs: bor1
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
Keywords: obesity, etiology, pathogenesis, treatment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- normal: body mass index: 19-24
- overweight: body mass index: 25-29
- obesity: body mass index: 30-40
- modbid obes: body mass index: over 40

SUMMARY:
According to our experimental experiences w hypothesized that blood boron levels may be corralated to body mass index.

DETAILED DESCRIPTION:
In the results of our experimental study on mices we revealed that low dose oral boric acid intake cause seriously body mas reducing. Although blood and urine analyses support high glucose, lipid and middle protein catabolisms, but the mechanism was unclear. There are some diseases according to blood elementary deficiencies, like hypothyroidi in hypoiyodinemia, hiperparathyroidi in hypocalcemia, etc. We hypothesised that hypoboronemia may be corralated to body mass index level.

ELIGIBILITY:
Inclusion Criteria:

* body mas index levels in over 19 peoples

Exclusion Criteria:

* known chronic, morbid and malign diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal: 19-24 Overweight: 25-29 Obes: 30-40 Morbid Obes: >40
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
blood boron level | 6 months
  blood boron levels will be measured cantitatively

SECONDARY OUTCOMES:
body mass index | 6 months
  body mass index levels will be evaluated with blood boron levels

CONTACTS AND LOCATIONS:
Overall Officials: adnan yuksel, prof, Study Chair — rector
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Aysan E, Bektas H, Ersoz F, Sari S, Kaygusuz A. A novel colonic anastomosis technique involving fixed polyglycolic acid mesh. Int J Clin Exp Med. 2010 Oct 24;3(4):341-6. PMID 21072268